CLINICAL TRIAL: NCT02505308
Title: Defining the Molecular and Physiological Mechanisms of Pancreatic Islet Cell Dysfunction Which Lead to Type 2 Diabetes (DIabetes VAriants)
Brief Title: Defining the Molecular and Physiological Mechanisms of Pancreatic Islet Cell Dysfunction Which Lead to Type 2 Diabetes
Acronym: DIVA-Exeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); University of Oxford (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CRF 172; 1507116 (Other: Royal Devon & Exeter NHS Foundation Trust R&D); 18599 (Other: UKCLRN)
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus
Keywords: insulin; proinsulin; genotype; beta cells; physiology; genetics; pathogenesis; rare variants; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Insulin-Dependent, 2; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DIVA-1 CCND2 (Experimental): Individuals carrying a genetic change in the CCND2 gene and controls matched for gender, age and BMI. Participants will undergo the Glucose-Potentiated Arginine-Induced Insulin Secretion (GPAIS) test plus optional faecal elastase measurement. Case/control status will be unblinded at analysis.
  Interventions: Other: Glucose-Potentiated Arginine-Induced Insulin Secretion
- DIVA-2 Low Risk of Diabetes (Experimental): Individuals carrying the fewest genetic risk alleles for diabetes and controls carrying the average number of genetic risk alleles, matched for gender, age and BMI. Participants will undergo the Glucose-Potentiated Arginine-Induced Insulin Secretion (GPAIS) test plus optional faecal elastase measurement. Case/control status will be unblinded at analysis.
  Interventions: Other: Glucose-Potentiated Arginine-Induced Insulin Secretion

INTERVENTIONS:
Other: Glucose-Potentiated Arginine-Induced Insulin Secretion — Intravenous catheters are inserted into antecubital veins in both arms. One arm is used for infusion of glucose/amino acid (Arginine). The other arm is used for intermittent sampling.
  Other Names: GPAIS test

SUMMARY:
Defects in insulin secretion are central to the pathogenesis of type 2 diabetes (T2D) but the molecular basis and physiological consequences of those defects are poorly understood, impeding efforts to develop novel therapeutic approaches. Key questions remain unanswered, such as the extent to which T2D-associated islet dysfunction reflects endogenous defects in beta-cell mass or function, as opposed to disruption of external factors impinging on the beta-cells, such as incretins.

Recently the investigators have identified several genetic variations (DNA changes) associated with the production and processing of insulin in non-diabetic individuals and now aim to explore in more detail the role of these genetic variations. Utilising a "recruit by genotype" approach, they will identify individuals with and without genetic variants of interest from existing databases of research volunteers. The investigators will collect detailed medical history and measurements, fasted and stimulated blood samples for the profiling of insulin-related hormones and metabolites. The resulting genetic and non-genetic data will be used to improve understanding of the role of genetic variation on insulin secretion and sensitivity defects that lead to the development of T2D.

DETAILED DESCRIPTION:
Introduction:

Working with collaborators as part of ongoing genetic studies, the investigators have identified several genetic variations (DNA changes) associated with the production of and processing of insulin and are trying to understand how these genetic variations cause differences in people's ability to produce or process insulin. Their findings will lead to an improved understanding of how the pancreas produces and processes insulin after a meal and will help to improve understanding of why some people develop diabetes and some people do not, despite similar levels of obesity. This question is of great public health significance because it is unlikely that the prevalence of obesity will fall dramatically in the foreseeable future.

The investigators would like to test the hypothesis that individuals carrying different genetic variations have different abilities to produce or process insulin. They will test the consequences of these genetic variations when the pancreas has to produce insulin in response to a meal or components of a meal, such as sugar or amino acids.

Study design:

This is a prospective "recruit by genotype" cohort study that will test the role of several genetic variants (or combinations of variants) over a 4 year period (late 2014 to late 2018). The genetic variants will be chosen if there is strong evidence that they have a role in the pancreas and on insulin secretion. Each genetic variant will involve a different set of research volunteers and a slightly different set of tests. Participants will be blinded to their genetic variant status. Some genetic variants will be identified during the next 4 years so it is not possible to define at the outset a detailed methodology for all cohorts to be studied. This protocol has therefore been written to describe a core protocol relevant to the whole study, with appendices to describe specific cohorts within the study. Since the general management and ethical issues are overarching, as new genetic variants are identified over the 4 year study period, cohort-specific appendices will be added as major amendments, rather than submitting each cohort as a separate ethics application. The procedure for recruitment and testing of each set of research volunteers will be the same except for a component that will be outlined in cohort-specific appendices.

Study participants:

All participants will be identified from existing research cohorts managed by the NIHR Exeter Research Facility (Exeter CRF) and/or the Oxford Biobank (OBB) and recruitment will be facilitated within the Exeter CRF and/or Oxford Centre for Diabetes, Endocrinology and Medicine (OCDEM). Individuals will be identified with the variant of interest or as gender, age and BMI matched controls. All potential participants will be 'blinded' by a Data Manager so that the study team does not know which participants have the variant and which are controls. They will be invited into the study by letter, and provided with the study information sheet and study team contact details. A member of the study team will contact them within 2-3 weeks to determine whether they are interested in participating, to offer them greater explanation of what the study entails, and to check their eligibility. If they agree to take part, verbal consent for a fasted visit will be sought and an appointment will be made and confirmed in writing/by email.

Identifying genetic variation:

Measuring the genetic factors in these individuals is an ongoing process that involves routine lab measures using the single existing DNA sample that the volunteers provided during their participation in the Exeter 10000 Project/OBB. As of June 2014, in Exeter 94 genetic variants (aka DNA changes) have been measured in 5600 EXTEND volunteers and 800,000 genetic variants in a subset of 1700 EXTEND volunteers. During the course of the next 4 years, the genetic measures will be extended to all participants (up to 10,000) and all variants (800,000+). These data will be returned to the EXTEND/OBB database as required.

Individuals identified with a genetic variation of interest will be invited to participate (30-50, dependent on the associated specific tests) together with a similar number of gender, age, and BMI matched control individuals without the variation of interest. The definition of matching will be same sex, age +/- 1 year, and BMI within 1 kgm2 unit but these ranges may be broadened if not enough individuals are available in the tighter definition.

Visit procedure:

All participants will be asked to fast overnight (from 10 pm the night before), avoid strenuous exercise and smoking for 24 hours prior to attending a morning visit at the Exeter CRF/OCDEM (approx 2-4 hours depending on test choice). Participants will be asked to sign a written consent form prior to any data collection or test. Patients who lack capacity to consent will not be recruited. Participants will be given the opportunity to contact a member of the research team to discuss the project in more detail if desired. All participants will be informed of the nature and purpose of the study, its requirements and possible hazards, and their rights to withdraw at any time from the study without prejudice and without jeopardy to any future clinical care.

All participants will undergo core data collection, measurements and provide fasted and stimulated blood samples. A cohort of participants may be asked to return for a second visit to undergo a further test to provide comparison measures. Test choice depends on the genetic variation being studied - detailed in cohort-specific appendices.

Core data collection, measurements and samples for all participants - approx. 1 hour Anthropometry: data, including Height (m), Weight (Kg), Waist (cm) and Hip (cm) circumference, will be recorded.

Medical history: including current medications and lifestyle information (smoking/alcohol).

BOD POD: Participants will be asked to have their fat mass measured by BOD POD. This non-invasive technique provides a more accurate measure of fat mass compared to bioimpedence measures, or measures of height and weight. Participants that opt out of this test will not be excluded from the study.

Detailed body composition measures will be obtained using the Body Composition Tracking System. This briefly comprises a BOD POD machine, electronic scales, and a computer. It uses the principles of body densitometry (measuring mass and volume) to calculate the participant's percentage and absolute amounts of fat and fat free mass. Participants will be asked to wear minimal clothing (e.g. swimming costume) and a close fitting swim hat. They stand on the electric scales to record their weight which is then calibrated with the BOD POD. Participants are asked to sit inside the BOD POD for up to 1 minute at a time (max 3 times). The computer will then analyze and generate the results.

Blood samples:

A small cannula (thin plastic tube) will be inserted into a vein, following standard clinical practice to minimise any potential trauma from repeat blood sampling.

Fasted samples will be obtained for baseline measures (including routine glucose and lipid measurement), DNA, plasma, and serum, for storage and future batched analysis including measures of glucose and insulin and other markers of interest.

Stimulated blood samples will be obtained from all participants. The choice of stimulation agent will be dependent on the specific genetic variation under study. At the end of the test period, the cannula will be removed and the participant will be offered breakfast/refreshments.

Definitions of the genotypes of interest and details of the visit(s) are provided in the protocol's cohort-specific appendices. In addition to the core data collection, measurements and fasted samples, each cohort will undertake up to two of the tests described below.

A: Glucose-Potentiated Arginine-Induced Insulin secretion (GPAIS) - approx. 1½ hrs Rationale. This test is designed primarily to test the maximum insulin secretion capacity of a participant's beta cells. It provides the best available surrogate for beta cell mass, as opposed to beta cell function (Kahn 2008) and will therefore help to improve understanding of the mechanisms of how chosen genetic variants influence risk of diabetes. It has recently been shown to correlate well with the number of (autologous) islets transplanted into pancreatitis patients following pancreatectomy. In dogs and non-human primates it correlates well with % beta cell mass (reviewed in Kahn 3). The test is based on the well-described (Kahn 2008; Larsson & Ahren 1998) principle that a non-glucose secretagogue, such as the amino acid arginine, will produce greater insulin response when potentiated by high glucose levels, with the combined stimulus producing a near maximal beta cell response.

The GPAIS test involves 5 stages:

1. Set up. Intravenous catheters will be inserted into antecubital veins in both arms. One arm will be used for infusion of glucose/amino acid, and the other arm for intermittent sampling. Blood glucose concentration will be monitored with regular YSI measures throughout the test.
2. AIRarg (acute insulin response to arginine). Baseline samples will be taken at -2 and -0 min. A maximally stimulating bolus dose of arginine hydrochloride (5 g) will then be injected intravenously for 45 s. Samples will be collected at +2, +3, +4 and +5 min.
3. Acute insulin response to intravenous glucose (unvalidated measure of acute insulin response to intravenous glucose AIRglucose). Next a high-speed (900 ml/hr) 20% glucose infusion over 10-25 minutes will be commenced (total volume infused up to 410 ml). Samples will be collected at -5, -2 min (before starting the high speed infusion) and then at 2 minute intervals for 10 minutes following the start of the glucose infusion.
4. AIRMAXarg. When the glucose levels have reached 20mmol/L (or after 25 mins max), repeat baseline samples will be taken, the glucose infusion lowered to 300ml/hr and a second arginine hydrochloride (5 g) bolus will be injected, followed by final +2, +3, +4 and +5 min samples.
5. Recovery and monitoring of glucose and insulin as participant's glucose levels return to baseline. Samples for glucose and insulin will be collected every 10 minutes for 50 minutes after the end of the AIRMAXarg test to monitor the participant's recovery and provide a measure of insulin sensitivity. Blood sugar will be monitored with regular YSI measures until the participant's blood sugar returns to a safe level. The participant will be given a light lunch at the end of this period.

Samples: at all time points insulin and glucose will be measured. Spare aliquots will be saved and stored at -80oC for potential additional analysis, such as glucagon and C-peptide.

B: Intravenous Glucose Tolerance Test (IGTT aka IVGTT) - approx. 30 minutes Rationale. This test is an accepted, standard measure of first phase insulin secretion that does not involve the neurohormonal (incretin) and absorption effects of an oral glucose challenge.

C: Oral Glucose Tolerance Test (OGTT) - approx. 2.5 hrs Rationale. This test is an accepted, standard measure of insulin secretion and absorption effects of an oral glucose challenge.

D: Stool sample for faecal elastase measurement Rationale. This will test the hypothesis that the genetic polymorphism may influence exocrine pancreatic function in addition to pancreatic endocrine function.

The participant will be provided with a specimen container, prepaid padded envelope, transport container, and instructions to collect and post a faecal sample for analysis. Provision of a faecal sample will be optional and will not be essential for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: Adult, age 16-75 inclusive
* Ethnicity: Reflective of local demographic
* Mental capacity: Capacity to consent

Exclusion Criteria:

* Demographics: <16 and >75 years old
* Medical history: Bariatric surgery; history of recent significant weight loss (>10% of weight in last year); known cardiovascular disease (previous myocardial infarction, stroke, angina or heart failure); glucose-galactose malabsorption syndrome; allergy to corn (maize)
* Medications: Currently prescribed glucose-lowering medication, oral/IV corticosteroid treatment or loop diuretics (furosemide, bumetanide)
* Mental capacity: Incapacity to consent

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Maximal Insulin Secretion (composite measure) following formal stimulation (GPAIS) test | Within 12 months of recruitment date of final participant
  Maximal insulin secretion will be assessed using composite measures of insulin, proinsulin, C-peptide, glucose, etc., from biological samples.

SECONDARY OUTCOMES:
Faecal elastase | Within 12 months of recruitment date of final participant
  Faecal elastase as a secondary measure of pancreas size

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Frayling (Prof), PhD, Principal Investigator — University of Exeter
Locations (2):
- United Kingdom (2):
  - University of Exeter, Exeter, Devon
  - University of Oxford, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahn SE, Carr DB, Faulenbach MV, Utzschneider KM. An examination of beta-cell function measures and their potential use for estimating beta-cell mass. Diabetes Obes Metab. 2008 Nov;10 Suppl 4:63-76. doi: 10.1111/j.1463-1326.2008.00945.x. PMID 18834434
- [Background] Larsson H, Ahren B. Glucose-dependent arginine stimulation test for characterization of islet function: studies on reproducibility and priming effect of arginine. Diabetologia. 1998 Jul;41(7):772-7. doi: 10.1007/s001250050986. PMID 9686917